CLINICAL TRIAL: NCT00346632
Title: Phase I Safety, Pharmacokinetic, and Pharmacodynamic Study of KW-2449 in Acute Leukemias (AML), Myelodysplastic Syndromes (MDS), and Chronic Myelogenous Leukemia (CML)
Brief Title: An Ascending Dose Study of KW-2449 in Acute Leukemias, Myelodysplastic Syndromes, and Chronic Myelogenous Leukemia
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Terminated due to suboptimal dosing schedule
Sponsor: Kyowa Kirin, Inc. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2449-US-001
Record Dates: First submitted 2006-06-28; First posted 2006-06-30 (Estimated); Results first posted 2016-08-12 (Estimated); Last update posted 2024-05-17 (Actual); Status verified 2024-04

CONDITIONS: Acute Myelogenous Leukemia; Acute Lymphoblastic Leukemia; Myelodysplastic Syndromes; Chronic Myelogenous Leukemia
Keywords: AML; ALL; MDS; CML; Kinase Inhibitor
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Myelodysplastic Syndromes; Leukemia, Myelogenous, Chronic, BCR-ABL Positive | interventions — KW 2449

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- KW-2449 (Experimental): Treatment with ascending doses of KW-2449
  Interventions: Drug: KW-2449

INTERVENTIONS:
Drug: KW-2449 — Sequential ascending oral doses of KW-2449 given for 14 or 28 days (modified by protocol amendment to only 14 days dosing).

SUMMARY:
Non-randomized, open, dose ranging and dose scheduling study of ascending doses of KW-2449 in subjects with AML, ALL, MDS and CML.

DETAILED DESCRIPTION:
This is a Phase I open-label dose escalation study of KW-2449 in subjects with acute leukemias, high risk MDS, and CML who are not candidates for approved therapy. Over an 18-month period, the investigative sites collectively will enroll up to a total of 96 subjects. Subjects will be enrolled sequentially into 1 of 7 dose groups to evaluate 2 dosing schedules (Arm A = 14 consecutive days of dosing followed by a 7-28 day rest period as determined by recovery from any acute hematologic and non-hematologic toxicities, or Arm B = 28 consecutive days of dosing followed by a 7-28 day rest period, as determined by recovery from any acute hematologic and non-hematologic toxicities). The safety of a dose level in Arm A (14-day dosing regimen) will be established prior to enrollment of subjects in the same dose level in Arm B (28-day dosing regimen).

In April 2007 the protocol was amended to discontinue Arm B (28 consecutive days of dosing). The protocol will continue as planned for Arm A (14 days of consecutive dosing).

Enrollment will proceed until a maximum tolerated dose (MTD) has been established for each study Arm. Once the MTD has been reached, 12 additional subjects, with 1 or more of the hematologic conditions included in this study, may be enrolled at the MTD as an expanded safety cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed diagnosis of:

   * AML (including APL refractory to all-trans retinoic acid and arsenic) that has relapsed or was not responsive to prior chemotherapy;
   * Relapsed/refractory ALL;
   * CML that has failed to respond or has lost a response to imatinib; and
   * Advanced MDS (INT-2 and High risk by IPSS) with failure or intolerance to approved therapy.
2. ECOG Performance Status score of 0, 1, or 2;
3. Male or female, at least 18 years of age;
4. Signed written informed consent;
5. Serum creatinine ≤ 2.0 mg/dL;
6. Serum SGOT (AST) and SGPT (ALT) ≤ 5x ULN; serum bilirubin ≤ 2 mg/dL (serum bilirubin may be ≤ 3.0 mg/dL in any subject with Gilbert's Syndrome); and
7. For females of childbearing potential, a negative serum pregnancy test. Subjects, of childbearing potential, must use an Investigator-approved method of birth control.

Exclusion Criteria:

1. Candidates for approved therapies;
2. Concomitant treatment with any investigational agent, chemotherapy, radiotherapy, or immunotherapy;
3. Active CNS leukemia;
4. Previous or concurrent malignancy except noninvasive non-melanomatous skin cancer, in situ carcinoma of the cervix, or other solid tumor treated curatively, and without evidence of recurrence for at least 2 years prior to study entry;
5. Uncontrolled systemic infection (viral, bacterial, or fungal);
6. Uncontrollable disseminated intravascular coagulation;
7. Major surgery within the 28 days preceding the first dose KW-2449;
8. Radiotherapy, or lack of recovery of any radiotherapy-related acute toxicity, within the 28 days preceding the first dose KW-2449;
9. Treatment with systemic therapy for the underlying hematologic condition, or lack of recovery of toxicity from such treatment, within 28 days of the first dose of KW-2449, with the following exceptions: hydroxyurea for treatment of hyperleukocytosis (discontinued for at least 48 hours prior to the first dose of KW-2449); imatinib (discontinued for at least 48 hours prior to the first dose of KW-2449); and interferon (discontinued for at least 7 days prior to the first dose of KW-2449);
10. Treatment with any other investigational agent, or lack of recovery of toxicity from such treatment, within the 28 days preceding the first dose of KW-2449;
11. Positive serology for HIV;
12. Clinically significant cardiac dysfunction (New York Heart Association Class 3 or 4) at the time of screening, or a history of myocardial infarction or heart failure within 3 months preceding the first dose of KW-2449;
13. Any evidence of chronic Graft versus Host Disease;
14. Active autoimmune disease requiring immunosuppressive therapy;
15. Female subjects who are pregnant or breast feeding;
16. Subjects of childbearing potential, unwilling to use an approved, effective means of contraception in accordance with the institution's standards;
17. Known current drug or alcohol abuse;
18. Other severe, acute, or chronic medical or psychiatric condition, or laboratory abnormality that may compromise the safety of the subject during the study, affect the subject's ability to complete the study, or interfere with interpretation of study results; or
19. For any reason is judged by the Investigator to be inappropriate for study participation, including an inability to communicate or cooperate with the Investigator.
20. Hematopoietic growth factors (i.e., such as erythropoietin or darbepoetin alpha, filgrastim [granulocyte colony-stimulating factor {G-CSF }], sargramostim [granulocyte-macrophage colony-stimulating factor {GM-CSF}], or other thrombopoietic agents) and corticosteroids within 14 days of study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2006-06; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matt Fujimori, MD, Study Director — Kyowa Kirin, Inc.
Locations (4):
- United States (4):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Contact Kyowa, Princeton, New Jersey
  - Weill Cornell/New York Presbyterian Hospital, New York, New York
  - M.D. Anderson Cancer Center, Houston, Texas

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Pratz KW, Cortes J, Roboz GJ, Rao N, Arowojolu O, Stine A, Shiotsu Y, Shudo A, Akinaga S, Small D, Karp JE, Levis M. A pharmacodynamic study of the FLT3 inhibitor KW-2449 yields insight into the basis for clinical response. Blood. 2009 Apr 23;113(17):3938-46. doi: 10.1182/blood-2008-09-177030. Epub 2008 Nov 24. PMID 19029442

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Four study centers in the US
Groups:
- 25 mg/Day KW-2449 14-day Regimen (Arm A); 50 mg/Day KW-2449 14-day Regimen (Arm A); 100 mg/Day KW-2449 14-day Regimen (Arm A); 200 mg/Day KW-2449 14-day Regimen (Arm A); 300 mg/Day KW-2449 14-day Regimen (Arm A); 400 mg/Day KW-2449 14-day Regimen (Arm A); 500 mg/Day KW-2449 14-day Regimen (Arm A): Arm A has sequential ascending oral doses of KW-2449 given for 14-day cycles
- 25 mg/Day KW-2449 28-day Regimen (Arm B); 50 mg/Day KW-2449 28-day Regimen (Arm B); 100 mg/Day KW-2449 28-day Regimen (Arm B): Arm B has sequential ascending oral doses of KW-2449 given for 28-day cycles
Period: Overall Study
Arm/Group | 25 mg/Day KW-2449 14-day Regimen (Arm A) | 50 mg/Day KW-2449 14-day Regimen (Arm A) | 100 mg/Day KW-2449 14-day Regimen (Arm A) | 200 mg/Day KW-2449 14-day Regimen (Arm A) | 300 mg/Day KW-2449 14-day Regimen (Arm A) | 400 mg/Day KW-2449 14-day Regimen (Arm A) | 500 mg/Day KW-2449 14-day Regimen (Arm A) | 25 mg/Day KW-2449 28-day Regimen (Arm B) | 50 mg/Day KW-2449 28-day Regimen (Arm B) | 100 mg/Day KW-2449 28-day Regimen (Arm B)
Started | 3 | 3 | 6 | 3 | 4 | 2 | 5 | 4 | 4 | 3
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 3 | 3 | 6 | 3 | 4 | 2 | 5 | 4 | 4 | 3
Not completed — Progressive Disease | 2 | 2 | 4 | 3 | 3 | 1 | 2 | 2 | 2 | 2
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 1 | 1 | 1 | 0 | 0 | 0
Not completed — Death | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Not completed — Switched to alternative treatment | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Not Stated | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm A: KW-2449 14-day Regimen: Sequential ascending oral doses of KW-2449 given for 14-day cycles
- Arm B: KW-2449 28-day Regimen: Sequential ascending oral doses of KW-2449 given for 28-day cycles
- Total: Total of all reporting groups
Arm/Group | Arm A: KW-2449 14-day Regimen | Arm B: KW-2449 28-day Regimen | Total
Number analyzed (Participants) | 26 | 11 | 37
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 18 | 5 | 23
  >=65 years | 8 | 6 | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.4 (15.48) | 62.1 (17.22) | 61.6 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 6 | 21
  Male | 11 | 5 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 1 | 3
  White | 23 | 10 | 33
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 26 | 11 | 37

OUTCOME MEASURES:

1. Primary Outcome: Safety of KW-2449 - Number of Participants With Treatment-related Adverse Events (TEAEs) as Assessed by NCI-CTCAE v3.0
Description: In addition to the number of TEAEs, the number of serious TEAEs, the number of related TEAEs, the number of Grade 3-4 TEAEs, and the number of subjects who died or discontinued due to TEAEs were also assessed. The maximally tolerated dose (MTD) was also to be determined, but it was not actually reached in either arm.
Time Frame: Baseline up to Cycle 2, Day 1
Measure: Number; unit: participants
Groups:
- Arm A - 25 mg/Day: KW2449-001 25 mg/day (Treatment Arm A)
- Arm A - 50 mg/Day: KW2449-001 50 mg/day (Treatment Arm A)
- Arm A - 100 mg/Day: KW2449-001 100 mg/day (Treatment Arm A)
- Arm A - 200 mg/Day: KW2449-001 200 mg/day (Treatment Arm A)
- Arm A - 300 mg/Day: KW2449-001 300 mg/day (Treatment Arm A)
- Arm A - 400 mg/Day: KW2449-001 400 mg/day (Treatment Arm A)
- Arm A - 500 mg/Day: KW2449-001 500 mg/day (Treatment Arm A)
- Arm A - Total: Total Patients in Treatment Arm A
- Arm B - 25 mg/Day: KW2449-001 25 mg/day (Treatment Arm B)
- Arm B - 50 mg/Day: KW2449-001 50 mg/day (Treatment Arm B)
- Arm B - 100 mg/Day: KW2449-001 100 mg/day (Treatment Arm B)
- Arm B - Total: Total Patients in Treatment Arm B
Arm/Group | Arm A - 25 mg/Day | Arm A - 50 mg/Day | Arm A - 100 mg/Day | Arm A - 200 mg/Day | Arm A - 300 mg/Day | Arm A - 400 mg/Day | Arm A - 500 mg/Day | Arm A - Total | Arm B - 25 mg/Day | Arm B - 50 mg/Day | Arm B - 100 mg/Day | Arm B - Total
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 4 | 2 | 5 | 26 | 4 | 4 | 3 | 11
participants
  Subjects with any TEAE | 3 | 3 | 6 | 3 | 4 | 2 | 5 | 26 | 4 | 4 | 3 | 11
  Subjects with any serious TEAE | 2 | 2 | 5 | 2 | 4 | 1 | 3 | 19 | 2 | 3 | 3 | 8
  Subjects with TEAE related to study drug | 1 | 3 | 6 | 3 | 4 | 2 | 3 | 22 | 3 | 3 | 3 | 9
  Subjects with TEAE of Grade 3 or above | 2 | 2 | 6 | 2 | 4 | 2 | 3 | 21 | 1 | 3 | 3 | 7
  Subjects who discontinued the study due to TEA | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Subjects who died | 1 | 0 | 5 | 1 | 3 | 0 | 1 | 11 | 0 | 1 | 0 | 1

2. Secondary Outcome: Observed Peak Plasma Concentration (Cmax)
Time Frame: Days 1 and 14 (and Day 28 for Arm B) of Cycle 1
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Arm A - 25 mg/Day: Day 1; Arm A - 25 mg/Day: Day 14: KW2449-001 25 mg/day (Treatment Arm A)
- Arm A - 50 mg/Day: Day 1; Arm A - 50 mg/Day: Day 14: KW2449-001 50 mg/day (Treatment Arm A)
- Arm A - 100 mg/Day: Day 1; Arm A - 100 mg/Day: Day 14; Arm B - 100 mg.Day: Day 1: KW2449-001 100 mg/day (Treatment Arm A)
- Arm A - 200 mg/Day: Day 1; Arm A - 200 mg/Day: Day 14: KW2449-001 200 mg/day (Treatment Arm A)
- Arm A - 300 mg/Day: Day 1; Arm A - 300 mg/Day: Day 14: KW2449-001 300 mg/day (Treatment Arm A)
- Arm A - 400 mg/Day: Day 1; Arm A - 400 mg/Day: Day 14: KW2449-001 400 mg/day (Treatment Arm A)
- Arm A - 500 mg/Day: Day 1; Arm A - 500 mg/Day: Day 14: KW2449-001 500 mg/day (Treatment Arm A)
- Arm B - 25 mg/Day: Day 1; Arm B - 25 mg/Day: Day 14; Arm B - 25 mg/Day: Day 28: KW2449-001 25 mg/day (Treatment Arm B)
- Arm B - 50 mg/Day: Day 1; Arm B - 50 mg/Day: Day 14; Arm B - 50 mg/Day: Day 28: KW2449-001 50 mg/day (Treatment Arm B)
- Arm B - 100 mg/Day: Day 14; Arm B - 100 mg/Day: Day 28: KW2449-001 100 mg/day (Treatment Arm B)
Arm/Group | Arm A - 25 mg/Day: Day 1 | Arm A - 25 mg/Day: Day 14 | Arm A - 50 mg/Day: Day 1 | Arm A - 50 mg/Day: Day 14 | Arm A - 100 mg/Day: Day 1 | Arm A - 100 mg/Day: Day 14 | Arm A - 200 mg/Day: Day 1 | Arm A - 200 mg/Day: Day 14 | Arm A - 300 mg/Day: Day 1 | Arm A - 300 mg/Day: Day 14 | Arm A - 400 mg/Day: Day 1 | Arm A - 400 mg/Day: Day 14 | Arm A - 500 mg/Day: Day 1 | Arm A - 500 mg/Day: Day 14 | Arm B - 25 mg/Day: Day 1 | Arm B - 25 mg/Day: Day 14 | Arm B - 25 mg/Day: Day 28 | Arm B - 50 mg/Day: Day 1 | Arm B - 50 mg/Day: Day 14 | Arm B - 50 mg/Day: Day 28 | Arm B - 100 mg.Day: Day 1 | Arm B - 100 mg/Day: Day 14 | Arm B - 100 mg/Day: Day 28
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 3 | 3 | 4 | 4 | 2 | 2 | 5 | 5 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 3 | 3
ng/mL | 6.35 (0.754) | 7.94 (3.06) | 10.5 (3.49) | 18.6 (3.10) | 34.4 (15.7) | 38.8 (16.1) | 31.3 (17.8) | 83.7 (97.4) | 97.5 (18.6) | 147 (77.1) | 151 (52.3) | 198 (23.3) | 180 (125) | 371 (129) | 7.05 (4.85) | 8.39 (1.70) | 4.49 (1.97) | 8.20 (4.11) | 12.7 (4.73) | 15.6 (9.43) | 20.9 (9.66) | 36.3 (15.1) | 32.5 (24.6)

3. Secondary Outcome: Time to Peak Plasma Concentration (Tmax)
Time Frame: Days 1 and 14 (and Day 28 for Arm B) of Cycle 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Arm A - 25 mg/Day: Day 1 | Arm A - 25 mg/Day: Day 14 | Arm A - 50 mg/Day: Day 1 | Arm A - 50 mg/Day: Day 14 | Arm A - 100 mg/Day: Day 1 | Arm A - 100 mg/Day: Day 14 | Arm A - 200 mg/Day: Day 1 | Arm A - 200 mg/Day: Day 14 | Arm A - 300 mg/Day: Day 1 | Arm A - 300 mg/Day: Day 14 | Arm A - 400 mg/Day: Day 1 | Arm A - 400 mg/Day: Day 14 | Arm A - 500 mg/Day: Day 1 | Arm A - 500 mg/Day: Day 14 | Arm B - 25 mg/Day: Day 1 | Arm B - 25 mg/Day: Day 14 | Arm B - 25 mg/Day: Day 28 | Arm B - 50 mg/Day: Day 1 | Arm B - 50 mg/Day: Day 14 | Arm B - 50 mg/Day: Day 28 | Arm B - 100 mg.Day: Day 1 | Arm B - 100 mg/Day: Day 14 | Arm B - 100 mg/Day: Day 28
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 3 | 3 | 4 | 4 | 2 | 2 | 5 | 5 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 3 | 3
hours | 1.51 (0.508) | 1.83 (1.18) | 1.67 (0.577) | 2.06 (0.0962) | 1.31 (0.386) | 0.979 (0.728) | 2.97 (1.71) | 2.68 (1.36) | 1.67 (0.577) | 1.50 (0.707) | 2.00 (0.00) | 1.57 (0.613) | 2.27 (1.23) | 1.50 (0.707) | 2.27 (1.28) | 1.14 (0.177) | 1.33 (0.583) | 1.26 (0.506) | 1.26 (0.492) | 1.44 (0.509) | 1.34 (0.587) | 2.00 (1.73) | 1.54 (0.766)

4. Secondary Outcome: Area Under the Plasma Concentration-time Curve From 0 to Tau (AUC (0-tau, Tau is the Dosing Interval))
Time Frame: Days 1 and 14 (and Day 28 for Arm B) of Cycle 1
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Arm A - 25 mg/Day: Day 1 | Arm A - 25 mg/Day: Day 14 | Arm A - 50 mg/Day: Day 1 | Arm A - 50 mg/Day: Day 14 | Arm A - 100 mg/Day: Day 1 | Arm A - 100 mg/Day: Day 14 | Arm A - 200 mg/Day: Day 1 | Arm A - 200 mg/Day: Day 14 | Arm A - 300 mg/Day: Day 1 | Arm A - 300 mg/Day: Day 14 | Arm A - 400 mg/Day: Day 1 | Arm A - 400 mg/Day: Day 14 | Arm A - 500 mg/Day: Day 1 | Arm A - 500 mg/Day: Day 14 | Arm B - 25 mg/Day: Day 1 | Arm B - 25 mg/Day: Day 14 | Arm B - 25 mg/Day: Day 28 | Arm B - 50 mg/Day: Day 1 | Arm B - 50 mg/Day: Day 14 | Arm B - 50 mg/Day: Day 28 | Arm B - 100 mg.Day: Day 1 | Arm B - 100 mg/Day: Day 14 | Arm B - 100 mg/Day: Day 28
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 3 | 3 | 4 | 4 | 2 | 2 | 5 | 5 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 3 | 3
hr*ng/mL | 23.6 (8.56) | 30.9 (NA) — Data cannot be located. Study completed in 2008 and none of the people who worked on the study are still with the company | 46.7 (11.1) | 77.9 (29.7) | 138 (41.8) | 162 (28.7) | 173 (90.5) | 647 (665) | 428 (192) | 626 (310) | 647 (73.5) | 1060 (300) | 822 (463) | 1200 (180) | 38.0 (18.0) | 35.3 (8.76) | 28.8 (7.36) | 36.3 (18.1) | 58.7 (21.7) | 60.3 (23.6) | 107 (31.2) | 158 (58.8) | 147 (90.9)

5. Secondary Outcome: Terminal Half Life (t 1/2)
Time Frame: Days 1 and 14 (and Day 28 for Arm B) of Cycle 1
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Arm A - 25 mg/Day: Day 1 | Arm A - 25 mg/Day: Day 14 | Arm A - 50 mg/Day: Day 1 | Arm A - 50 mg/Day: Day 14 | Arm A - 100 mg/Day: Day 1 | Arm A - 100 mg/Day: Day 14 | Arm A - 200 mg/Day: Day 1 | Arm A - 200 mg/Day: Day 14 | Arm A - 300 mg/Day: Day 1 | Arm A - 300 mg/Day: Day 14 | Arm A - 400 mg/Day: Day 1 | Arm A - 400 mg/Day: Day 14 | Arm A - 500 mg/Day: Day 1 | Arm A - 500 mg/Day: Day 14 | Arm B - 25 mg/Day: Day 1 | Arm B - 25 mg/Day: Day 14 | Arm B - 25 mg/Day: Day 28 | Arm B - 50 mg/Day: Day 1 | Arm B - 50 mg/Day: Day 14 | Arm B - 50 mg/Day: Day 28 | Arm B - 100 mg.Day: Day 1 | Arm B - 100 mg/Day: Day 14 | Arm B - 100 mg/Day: Day 28
Number analyzed (Participants) | 3 | 3 | 3 | 3 | 6 | 6 | 3 | 3 | 4 | 4 | 2 | 2 | 5 | 5 | 4 | 4 | 4 | 4 | 4 | 4 | 3 | 3 | 3
hours | 2.96 (1.42) | 3.36 (NA) — Data cannot be located. Study completed in 2008 and none of the people who worked on the study are still with the company | 2.67 (0.435) | 3.26 (0.631) | 3.11 (0.310) | 2.80 (0.187) | 3.27 (NA) — Data cannot be located. Study completed in 2008 and none of the people who worked on the study are still with the company | 3.04 (0.715) | 2.48 (0.158) | 2.44 (0.149) | 2.42 (0.06) | 2.83 (0.0806) | 2.93 (1.01) | 2.47 (0.105) | 2.78 (0.108) | 3.00 (0.453) | 3.35 (0.443) | 3.90 (1.43) | 3.32 (0.383) | 3.88 (1.64) | 2.97 (0.471) | 3.90 (1.62) | 3.16 (NA) — Data cannot be located. Study completed in 2008 and none of the people who worked on the study are still with the company

6. Secondary Outcome: Accumulation Ratio (AUC 0-tau Day 14 or 28 / AUC 0-tau Day 1)
Time Frame: Day 1 and either Day 14 or Day 28 of Cycle 1
Measure: Mean (Standard Deviation); unit: Ratio of hr*ng/mL
Arm/Group | Arm A - 25 mg/Day: Day 14 | Arm A - 50 mg/Day: Day 14 | Arm A - 100 mg/Day: Day 14 | Arm A - 200 mg/Day: Day 14 | Arm A - 300 mg/Day: Day 14 | Arm A - 400 mg/Day: Day 14 | Arm A - 500 mg/Day: Day 14 | Arm B - 25 mg/Day: Day 14 | Arm B - 25 mg/Day: Day 28 | Arm B - 50 mg/Day: Day 14 | Arm B - 50 mg/Day: Day 28 | Arm B - 100 mg/Day: Day 14 | Arm B - 100 mg/Day: Day 28
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 4 | 2 | 5 | 4 | 4 | 4 | 4 | 3 | 3
Ratio of hr*ng/mL | 1.50 (NA) — Data cannot be located. Study completed in 2008 and none of the people who worked on the study are still with the company | 1.66 (0.389) | 1.50 (0.459) | 3.37 (1.45) | 1.28 (0.0271) | 1.68 (0.654) | 0.846 (NA) — Data cannot be located. Study completed in 2008 and none of the people who worked on the study are still with the company | 0.953 (0.181) | 0.906 (0.622) | 1.42 (0.331) | 1.44 (0.180) | 1.50 (0.187) | 1.60 (NA) — Data cannot be located. Study completed in 2008 and none of the people who worked on the study are still with the company

7. Secondary Outcome: Disease Response
Description: Disease response (i.e., complete or partial remission) based on standard criteria:
  Cheson BD, Bennett JM, Kopecky KJ, Buchner T, Willman CL, Estey EH, et al. Revised recommendations of the International Working Group for diagnosis, standardization of response criteria, treatment outcomes, and reporting standards for therapeutic trials in acute myeloid leukemia. J Clin Oncol. 2003 Dec 15;21(24):4642-4649.
  Cheson BD, Bennett JM, Kantarjian H, Pinto A, Schiffer CA, Nimer SD, et al. Report of an international working group to standardize response criteria for myelodysplastic syndromes. Blood. 2000 Dec 1;96(12):3671-3674.
  VHA Pharmacy Benefits Management Strategic Healthcare Group and the Medical Advisory Panel. Criteria for use of Imatinib Mesylate (Gleevec®) [updated March 2002; cited 2005 Nov 16]. Available from: http://www.pbm.va.gov/archive/imatinibcriteria.pdf
Time Frame: Day 14 (Arm A) or Day 28 (Arm B) for all cycles
Measure: Number; unit: number of responders
Arm/Group | Arm A - 25 mg/Day | Arm A - 50 mg/Day | Arm A - 100 mg/Day | Arm A - 200 mg/Day | Arm A - 300 mg/Day | Arm A - 400 mg/Day | Arm A - 500 mg/Day | Arm A - Total | Arm B - 25 mg/Day | Arm B - 50 mg/Day | Arm B - 100 mg/Day | Arm B - Total
Number analyzed (Participants) | 3 | 3 | 6 | 3 | 4 | 2 | 5 | 26 | 4 | 4 | 3 | 11
number of responders | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm A - 25 mg/Day | Arm A - 50 mg/Day | Arm A - 100 mg/Day | Arm A - 200 mg/Day | Arm A - 300 mg/Day | Arm A - 400 mg/Day | Arm A - 500 mg/Day | Arm A - Total | Arm B - 25 mg/Day | Arm B - 50 mg/Day | Arm B - 100 mg/Day | Arm B - Total
Serious Adverse Events (participants affected / at risk) | 2/3 | 2/3 | 5/6 | 2/3 | 4/4 | 1/2 | 3/5 | 19/26 | 2/4 | 3/4 | 3/3 | 8/11
Other Adverse Events (participants affected / at risk) | 3/3 | 3/3 | 6/6 | 3/3 | 4/4 | 2/2 | 5/5 | 26/26 | 4/4 | 4/4 | 3/3 | 11/11
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - 25 mg/Day (N=3) | Arm A - 50 mg/Day (N=3) | Arm A - 100 mg/Day (N=6) | Arm A - 200 mg/Day (N=3) | Arm A - 300 mg/Day (N=4) | Arm A - 400 mg/Day (N=2) | Arm A - 500 mg/Day (N=5) | Arm A - Total (N=26) | Arm B - 25 mg/Day (N=4) | Arm B - 50 mg/Day (N=4) | Arm B - 100 mg/Day (N=3) | Arm B - Total (N=11)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 8 (8) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Atrial flutter (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rectal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter related complication (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Disease progression (General disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Catheter related infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Escherichia sepsis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Localised infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (5) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
Pneumonia fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Haemoglobin decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Acute myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tumour lysis syndrome (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Brain stem haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subarachnoid haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure acute (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - 25 mg/Day (N=3) | Arm A - 50 mg/Day (N=3) | Arm A - 100 mg/Day (N=6) | Arm A - 200 mg/Day (N=3) | Arm A - 300 mg/Day (N=4) | Arm A - 400 mg/Day (N=2) | Arm A - 500 mg/Day (N=5) | Arm A - Total (N=26) | Arm B - 25 mg/Day (N=4) | Arm B - 50 mg/Day (N=4) | Arm B - 100 mg/Day (N=3) | Arm B - Total (N=11)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 1 (5) | 2 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (9) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhagic diathesis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Lymphadenopathy (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Splenomegaly (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Angina pectoris (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Bundle branch block right (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Palpitations (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ventricular extrasystoles (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Congenital jaw malformation (Congenital, familial and genetic disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ear haemorrhage (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ear pain (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Conjunctival hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eye pain (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Keratoconjunctivitis sicca (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Macular degeneration (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Ocular hyperaemia (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pupillary reflex impaired (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Scleral discolouration (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Visual disturbance (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vitreous floaters (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distension (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 1 (3) | 1 (1) | 1 (2) | 1 (4) | 0 (0) | 1 (1) | 5 (11) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Constipation (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 5 (6) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 3 (3) | 1 (2) | 2 (2) | 8 (10) | 1 (2) | 2 (3) | 2 (2) | 5 (7)
Dry mouth (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (2) | 2 (3)
Dysphagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Faecal incontinence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gastrointestinal inflammation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gingival bleeding (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Gingival pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Haemorrhoids (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Melaena (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 2 (2) | 2 (2) | 3 (3) | 3 (3) | 3 (7) | 1 (1) | 3 (3) | 17 (21) | 1 (2) | 2 (3) | 2 (2) | 5 (7)
Odynophagia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Oral mucosal petechiae (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Salivary gland enlargement (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue coated (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tongue disorder (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Toothache (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 2 (3) | 2 (2) | 2 (4) | 2 (2) | 2 (3) | 2 (3) | 14 (19) | 1 (1) | 2 (3) | 1 (1) | 4 (5)
Asthenia (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 3 (4) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Catheter site bruise (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Catheter site haemorrhage (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Catheter site oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Catheter site pain (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Catheter site related reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Chest pain (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chills (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Fatigue (General disorders) | 0 (0) | 2 (4) | 4 (4) | 0 (0) | 2 (2) | 1 (1) | 2 (3) | 11 (14) | 2 (4) | 1 (1) | 2 (6) | 5 (11)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Inflammation (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Injection site reaction (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Local swelling (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Localised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Malaise (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Mucosa vesicle (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nodule (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Oedema (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oedema peripheral (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 5 (5) | 1 (2) | 2 (5) | 2 (3) | 5 (10)
Pain (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (4) | 5 (7) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Hepatomegaly (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Portal vein thrombosis (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Catheter site infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cellulitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Enterococcal infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Herpes zoster (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Oral candidiasis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Otitis externa (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pneumonia fungal (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinusitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Subcutaneous abscess (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tooth abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 1 (3)
Tooth infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood alkaline phosphatase increased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood glucose increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Blood magnesium decreased (Investigations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Breath sounds abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cardiac murmur (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Electrocardiogram ST-T change (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Full blood count decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Heart sounds abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Spleen palpable (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Sputum abnormal (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight decreased (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Anorexia (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 2 (3) | 0 (0) | 3 (4)
Appetite disorder (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Gout (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hypermagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyperphosphataemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperuricaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (3) | 2 (3) | 0 (0) | 1 (2) | 0 (0) | 1 (1) | 6 (9) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 1 (1) | 3 (3)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Weight fluctuation (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (3) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 1 (1) | 6 (10) | 3 (3) | 1 (1) | 0 (0) | 4 (4)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 4 (4) | 0 (0) | 2 (3) | 0 (0) | 2 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Osteitis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 1 (1) | 1 (1) | 1 (1) | 8 (8) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sacral pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0) | 0 (0) | 1 (2) | 1 (2)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Coordination abnormal (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Drooling (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysarthria (Nervous system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dysgeusia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Facial palsy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 1 (2) | 3 (3) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Hemiparesis (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypoaesthesia (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Lethargy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Restless legs syndrome (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 1 (2)
Sensory disturbance (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Sinus headache (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Unresponsive to verbal stimuli (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Depressed mood (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Eating disorder (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Hallucination, visual (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (2) | 2 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 5 (6) | 0 (0) | 2 (2) | 1 (1) | 3 (3)
Micturition urgency (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Renal failure (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary hesitation (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pelvic pain (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (4) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 7 (9) | 2 (2) | 1 (1) | 1 (3) | 4 (6)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 3 (3)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased upper airway secretion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Laryngeal haemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2)
Pharyngeal erythema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rales (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (4) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Blood blister (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dermatitis exfoliative (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry skin (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 4 (4)
Erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Excoriation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Increased tendency to bruise (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Night sweats (Skin and subcutaneous tissue disorders) | 1 (2) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Palmar erythema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Periorbital oedema (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Petechiae (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Rash macular (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Rash pruritic (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin lesion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 2 (2)
Swelling face (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Hypertension (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 4 (4) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other